CLINICAL TRIAL: NCT01477788
Title: Prediction of Ovarian Malignancy, in the Presence of Sonographic Pelvic Mass Using Patient History, Sonographic Parameters and Serum Markers
Brief Title: Prediction of Ovarian Malignancy in the Presence of Sonographic Pelvic Mass
Status: Withdrawn | Type: Observational
Why Stopped: The researcher Left the organization
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Other Study IDs: EMC-0083-09
Record Dates: First submitted 2011-11-13; First posted 2011-11-23 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2011-11

CONDITIONS: Ovarian Neoplasm
Keywords: pelvic mass; ovarian mass; ultrasound; serum markers; ovarian malignancy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women, sonographic ovarian mass: women that will arrive to the sonographic unit of the gynecological department with the sonographic diagnosis of ovarian mass

SUMMARY:
The objective of the study is to create a test that will discriminate between malignant and benign ovarian mass that was diagnosed by ultrasound. The investigators will examine about 800 women and at the end of the study the investigators will combine data from the woman's history, the sonographic characters of the mass and serum biological markers along with the woman's outcome (which means - whether the mass was malignant, benign, or disappeared or remained constant with no intervention).

DETAILED DESCRIPTION:
Patients that arrive to the sonographic unit of the gynecological department with a diagnosis of ovarian mass will have a sonographic examination that include: Trans-vaginal +- trans-abdominal ultrasound with Doppler and three dimensional sonographic exam. anamnestic data will be collected and serum test for CA 125, HE4 and CEA. The management of the specific patient will be according to the department protocol, regardless the study data. The investigators will collect data about operation outcome and histological results of women that will be operated. Women that won't be operated on will be followed up every 6 months by the study team.

At the end of the study a statistical analysis will be made to create a sensitive and specific test for the prediction of malignancy in sonographic diagnosed ovarian mass.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred with sonographic diagnosis of pelvic mass

Exclusion Criteria:

* Pregnant women
* Known gynecologic malignancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the department's sonographic unit with diagnosis of adnexal or pelvic or ovarian mass
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The risk of malignancy in the presence of pelvic mass demonstrated by sonography. | Up to 2 months after recruiting and examining the last participant of the study
  Using a combination of the results of US examination, patient's history and serum markers to predict the risk of malignancy in women with pelvic mass demonstrated by sonography.

SECONDARY OUTCOMES:
number and kind of operative complications | within one month after operation
  Information about operative complications will be collected from the files of participants who were operated
Reasons for intervention | within one month after operation
  The reasons that led the treating physician to choose a surgical treatment will be collected from the files of the participants who were operated
operative finding and histologic results | within one month after operation
  The operative finding and histologic results will be collected from the files of the participants who were operated

CONTACTS AND LOCATIONS:
Overall Officials: yfat kadan, MD, Principal Investigator — Department of Ob/Gyn, Haemek medical center, Afula Israel
Locations (1):
- Sonographic unit, Department of Ob/Gyn, Haemek medical center, Afula, Israel